CLINICAL TRIAL: NCT06801704
Title: The Effects of Top Set Training in Combination With Power Training in Subjects With Parkinson's Disease
Brief Title: Top Set and Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20241248
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Top Set Resistance Training (Other): Participants will be in this group receiving the top set resistance training for up to 12 weeks.
  Interventions: Behavioral: Top Set Resistance Training
- Power Resistance Training (Other): Participants will be in this group receiving the power resistance training for up to 12 weeks.
  Interventions: Behavioral: Power Resistance Training

INTERVENTIONS:
Behavioral: Top Set Resistance Training — Participants will receive four warm-up sets at increasingly higher resistance, followed by three sets of eight repetitions per set on six resistance-training exercises. During training participants will be allowed 1-minute rests between sets. Participants will come in person for up to 12 weeks, twice per week, for approximately 45 minutes per day.
  Arms: Top Set Resistance Training
Behavioral: Power Resistance Training — Participants will receive a total of 24 in-person training sessions using three sets of eight repetitions per set on six power resistance-training exercises. During training participants will be allowed 1-minute rests between sets. Participants will come in person for up to 12 weeks, twice per week, for approximately 45 minutes per day.
  Arms: Power Resistance Training

SUMMARY:
This project will focus on improving power in adults with Parkinson's disease, since power is related to performance of daily activities and memory and decision making. The study will compare traditional power training, where the participant does all exercises as fast as possible to top set resistance training, where the participant does power training, but it is preceded by warm-up sets that progress in weight until the participant reaches 90% of the person's maximum strength. If the top set method is better than traditional power training, it could be more beneficial than existing methods in improving independence in adults with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Parkinson's disease
* Between the ages of 30-90 years of age
* A Hoehn and Yahr score of ≤3, which will be provided by the participant's medical provider within 1 year of the study's inception.

Exclusion Criteria:

* Uncontrolled cardiovascular disease that prevents participation in a training program
* Documented HIV infection or another immunodeficiency syndrome
* Other neuromuscular diseases besides Parkinson's disease
* Current musculoskeletal injury that prevents exercise.
* Having a pacemaker
* Pregnancy
* Incarcerated individuals
* Montreal Cognitive Assessment Score below 18

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in neuromuscular performance as measured by power production. | Baseline, 12 weeks
  This test measures the power a person can produce at maximal speed using a load of 50% of 1RM for the chest press and leg press. There are no minimum or maximum scores. The higher score indicates higher power. Power shows how fast a person can do work. The test typically takes about five minutes. Unit of measure is Watts.
Change in neuromuscular performance as measured by 1-repetition maximum (1RM | Baseline, 12 weeks
  Maximal load that can be lifted in one repetition (1RM) will be assessed for in both leg press and chest press exercises. The loads on the testing equipment will be increased over 5 to 7 testing sets. The persons 1RM will be the highest load the person can move through the range of motion of the exercise. There are no minimum or maximum scores for this test.
  The test typically takes 5 to 10 minutes. The higher the 1RM the stronger the person is.

SECONDARY OUTCOMES:
Change in the Speed of the Ten-Meter Walk Test. | Baseline, 12 weeks
  The ten-meter walk test will be used to assess gait velocity. The participants will be asked to walk as quickly as possible in a straight line on a 10-m course marked at 0, 2, 8 and 10 m. On verbal command, participants will start on the 0-m mark and stop when they cross the 10-m mark. The total time to ambulate from the 2-m mark to the 8-m mark (6 m total) will be timed to the hundreds of a second. Two trials will be performed, and the average will be documented in meters per second. Sixty-second recoveries will be provided between trials. Total time is 420 seconds.
Changes in Swing time of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be swing time. Swing time is how long it takes to swing the back foot forward to initiate a new step. The unit of measurement is seconds.
Changes in Stance Time of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be stance time. Stance time is the duration of the time between heel strike and toe off the same foot. The unit of measurement is seconds.
Changes in Double Support Time of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be double support time. Double support time is how long both feet are in contact with the ground. The unit of measurement is seconds.
Changes in Step Time of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be step time. Step time is how long one foot is in contact with the ground. The unit of measurement is seconds.
Changes in Cadence of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be cadence. Cadence is the number of steps per minute. The unit of measurement is steps per minute.
Changes in Stride Length of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be stride length. Stride length is the distance covered when a person takes two steps. The unit of measurement is meters.
Changes in Step Length of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be step length. Step length is the distance covered when a person takes one step. The unit of measurement is meters.
Changes in Speed of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. Gait speed is how fast a person walks. The unit of measurement is meters per second.
Changes in Stride Width of Gait. | Baseline, 12 weeks
  Movement analyses will be performed during the ten-meter walk test. Stride width is the side-to-side distance between the line of the two feet during gait. The measurement is in meters.
Change in Time for the Five Times Sit-to-Stand Test. | Baseline, 12 weeks
  The five-time sit-to-stand test will be used to assess functional lower body strength. The participant will sit with arms folded across the chest and the back against the chair. On a verbal command, the participant will stand up and sit down five times as quickly as possible. Timing begins at "Go" and ends when the buttocks touch the chair after the fifth repetition. One practice and two testing trials will be performed. Time will be measured in seconds.
Change in Distance of the Seated Medicine Ball Throw. | Baseline, 12 weeks
  For the Seated Medicine Ball Throw, subjects will sit in an armless chair with the back against the chair back, while holding the 6-pound medicine ball against the chest. Subjects will then throw the ball at a perceived 45° angle as far as possible. Subjects must complete at least three practice trials; however, subjects will be allowed more trials until comfortable with the testing procedure. Upon starting the official trial, subjects will complete three separate attempts at each varying medicine ball, to nine trials in total. Each of the three trials within a given medicine ball will be separated by a 1-minute rest. Distance will be measured in centimeters.
Changes in the Six-Minute Walk Test | Baseline, 12 weeks
  The object of the test is to walk as far as possible for six minutes. The subject will walk at a normal pace around a marked course for six minutes. The subject may stop to rest and begin again at will. The distance covered indicates aerobic fitness. The further a person walks, the better cardiovascular condition. The units are meters.
Change in the time required to complete the Timed Up-and-Go Test. | Baseline, 12 weeks
  Upon verbal cue, the subject stands up, walks around a cone placed three meters from the front edge of the chair, and then returns to a seated position as quickly as possible. Time is measured in seconds. The faster the person completes the test the better the dynamic balance.
Change in Muscle Thickness using Ultrasound. | Baseline, 12 weeks
  Three images will be taken in the longitudinal view in B-mode. Muscle thickness will be measured by drawing a perpendicular line from the deep to superficial aponeurosis at the thickest region of each muscle. The unit of measurement is centimeters.
Change in Muscle Quality using Gray Scale. | Baseline, 12 weeks
  Muscle quality will be measured through ultrasound using a Gray Scale. The black and white pixels correspond to arbitrary values of 0 (darker) to 255 (lighter), with darker colors indicting more muscle and lighter colors indicating more fat.
Changes in the Parkinson's Disease Questionnaire. | Baseline, 12 weeks
  The Parkinson's Disease Questionnaire-39 is a 39-item self-report questionnaire that assesses Parkinson's disease-specific health-related quality over the last month across the eight quality of life dimensions and specific dimensions of functioning and well-being. Each question is scored from 0-4 points, with lower scores reflecting better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No